CLINICAL TRIAL: NCT05184660
Title: The Use of a Wearable Data Input Device (Google Glass, Microsoft HoloLens or GoPro Like Camera Mounted to Eyewear) to Collect Drug Delivery Event Data
Brief Title: Smart Eyewear to Automatically Detect Drug Delivery Events
Status: Recruiting | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Kelly Michaelsen, Assistant Professor, School of Medicine, University of Washington
Other Study IDs: STUDY00010313
Record Dates: First submitted 2021-12-02; First posted 2022-01-11 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Smart Eyewear
Keywords: automatic detection; smart eyewear; drug delivery; drug administration; patient safety; anesthetic drug; anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project is designed as a prospective observational study of medication preparation and delivery using a novel wearable data input device to automate detection of drug delivery events in the anesthesia workspace at University of Washington Medical Center.

DETAILED DESCRIPTION:
Detailed Summary: The goal of this study is to devise a high-fidelity system that automatically collects data about anesthesia care, specifically drug preparation and delivery to the patient. We use a novel wearable data input device that collects computer processed images (video only, no audio) to determine details of the preparation and delivery of medications in the operating room. The wearable data input device is used by an anesthesia provider. The device collects computer processed images and in the anesthesia workspace, which will be used to develop machine learning algorithms that can automatically recognize drug administration events in order to automate medical record keeping in this environment.

Procedure: The principle investigator or a study coordinator will review the electronic operating room schedule to screen for potential data collection. The operating room team will be notified of the study the day prior to and day of data collection. The consented anesthesia provider will wear a point of view device to record drug preparation and drug delivery events in the operating room. Video recordings will be edited to remove Protected Health Information (PHI). Edited footage will then be annotated by volunteers on a computer vision learning tool website. The computer processed images will be then used to develop machine learning algorithms that can automatically recognize drug administration events.

Participants: The initial recruitment goal for the study is 10 nurse anesthetists recording 5 days each in the operating room. Nurse anesthetists are recruited as participants through word of mouth. If determined after data analysis that additional data needs to collected, additional anesthesia providers will be consented.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesia providers (attending anesthesiologist or certified registered nurse anesthetist) who work in an operating room at University of Washington Montlake Medical Center

Exclusion Criteria:

* Medical students and anesthesiology residents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anesthesia providers (attending anesthesiologist or certified registered nurse anesthetist) who work in an operating room at University of Washington Montlake Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Operating room footage | 8-10 hours
  Operating room footage of drug preparation and drug delivery events recorded by anesthesia provider using a point-of-view device.

SECONDARY OUTCOMES:
Computer vision toolkit | 8-10 hours
  A computer vision toolkit which can identify syringes and medications in the hand of a provider in near real time.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Michaelsen, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No